CLINICAL TRIAL: NCT04553913
Title: Proof-of-Concept: A Device to Determine Return of Sensation After a Regional Anesthetic Block
Brief Title: A Device to Determine Return of Sensation From Spinal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00067142
Record Dates: First submitted 2020-09-11; First posted 2020-09-18 (Actual); Results first posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Sensation Diminished, Pinprick
Keywords: nerve block; spinal block; local anesthetic; regional anesthesia
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: All participants will have the device placed in the recovery room to determine resolution of regional anesthetics.
Masking Description: There is no masking. The PACU nurse will know the patient has the device; the only thing that he/she will not know is when the patient pushed the button to turn off the device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- cooling device placed (Experimental): A basic medical grade cooling pad will be secured to the non operative leg. Intermittent coolness will be assessed and subject will inform recovery room staff when sensation returns.
  Interventions: Device: cooling device
- standard of care no intervention (No Intervention): Subjects in intervention arm will serve as their own control; standard nursing pinprick testing on the same (non-operative) thigh

INTERVENTIONS:
Device: cooling device — device placed on patient in recovery on non surgical side to determine resolution of spinal anesthetics.
  Arms: cooling device placed

SUMMARY:
Participation in this study will involve having a pad wrapped onto the subject's non-surgical leg to detect when sensation returns after spinal anesthetic and while in recovery room. The pad is part of an approved medical device, but which has been modified and will be used in an experimental way. The device will run cold water through the pad wrapped to the subject's leg. The subject will be asked to press a stop button when they feel the pad gets cold. Nurses in the recovery area will also be testing return of sensation using a standard technique and this will be compared to when the subject begins to feel the cold.

DETAILED DESCRIPTION:
Regional anesthesia investigators have always shown interest in measuring the specific duration of neuraxial or peripheral nerve blocks, and how variations in block technique or medications affect that duration. Although ostensibly a simple concept, there are many sensory modalities available for block testing (light touch, cold or hot temperature, pain, pressure, etc.) and there is no consensus in the anesthesia literature on how best to measure the duration of nerve block (. Sensory testing is repetitive, and must be practical and consistent. Pinprick and cold sensation are commonly employed, and these modalities share the same afferent fibers (C-delta) so there is close overlap in the sensory loss mapping after regional block. With respect to pinprick sensation there can be variability in the sharpness, pressure, and reproducibility of a pinprick test. Testing for cold sensation may be more consistent, using a controlled stimulus temperature and duration, and there are different methods of testing such as a cooled glass vial (5℃) or Rolltemp (25℃).

Testing for long-acting blocks overnight adds an additional challenge since it requires repetitive subject awakening for assessment, and the interval for testing is a compromise between test specificity and sleep disruption. Again, there is no consensus on the proper interval for testing recovery from regional block.

Cold therapy is a commonly applied modality following strenuous exercise or during recovery from extremity surgery, and is expected to reduce tissue damage and relieve pain. There is some evidence of benefit but little consensus on the optimum interval and duration of therapy, and there are many approved medical devices available for use.

This investigation proposes an adaptation of an approved cold therapy device to administer automated, periodic cold stimulus at a location made insensate by regional block. When the subject perceives cold at that site, they will press a stop switch to discontinue cooling which will also stop a timer and give an accurate duration of the time to recovery of sensation at that site.

The concept will be tested by comparing the duration measured to the standard measurement of recovery from nerve block (spinal) employed by post-anesthesia care unit (PACU) nurses who will use pinprick (toothpick) testing of lumbar dermatomes every thirty minutes. If the device shows acceptable agreement with standard block recovery testing, a follow-up study would be its evaluation for long-duration block testing as an alternative to research assistant repeated testing overnight.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-75 y/o and scheduled to undergo unilateral primary knee or hip arthroplasty under spinal anesthesia with bupivacaine, ropivacaine or tetracaine will be eligible.

Exclusion Criteria:

* Patients will be excluded if pre-block sensation is abnormal in the L3 dermatome of the non-operative leg (neuropathy), or if spinal anesthesia is not performed or is unsuccessful.
* They will also be excluded if sensation has already returned in the L3 dermatome on arrival to the PACU.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seiha Kim, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 subjects served as their own controls, so only 15 subjects total. Two methods were used to assess the return of sensation on the same side/same non-operative leg after spinal block at the same time
Groups:
- All Participants: 15 subjects served as their own controls; two methods were used to assess the return of sensation on the same side/same non-operative leg after spinal block at the same time
Period: Overall Study
Arm/Group | All Participants
Started | 15
Completed | 9
Not Completed | 6
Not completed — patient's block resolved prior to PACU | 1
Not completed — did not use the device properly | 5

BASELINE CHARACTERISTICS:
Groups:
- Overall Subject Numbers: Subjects in the experimental arm serve as their own control.
Arm/Group | Overall Subject Numbers
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Block Recovery Time (Device)
Description: Time to resolution of subarachnoid block (minutes from injection) will be measured for the device on the (non-operative) thigh.
Time Frame: Baseline, from injection and up to 4 hours after injection
Population: Applies to experimental site only.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cooling Device Placed
Number analyzed (Participants) | 9
minutes | 40.7 (33.32)

2. Primary Outcome: Block Recovery Time (Pinprick Test)
Description: Time to resolution of subarachnoid block (minutes from injection) will be measured for the standard nursing pinprick testing on the same (non-operative) thigh.
Time Frame: Baseline, from injection and up to 4 hours after injection
Population: this outcome applies to the standard of care site only
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard of Care no Intervention
Number analyzed (Participants) | 9
minutes | 3.3 (12.36)

3. Secondary Outcome: Device Temperature Consistency
Description: Percentage of time the temperature sensor displays the pad temperature between 40 and 50 degrees F for the duration of the application
Time Frame: 2 hours after baseline
Population: Data not collected for this outcome.
Arm/Group | Cooling Device Placed
Number analyzed (Participants) | 0

4. Secondary Outcome: Cooling Pad Temperature (°F) at Stop Switch Activation
Time Frame: 2 hours after baseline
Population: applies only to experimental site group
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Cooling Device Placed
Number analyzed (Participants) | 9
degrees Fahrenheit | 53.9 (5.6)

ADVERSE EVENTS:
Time Frame: from baseline through completion of study, an average of four hours
Groups:
- All Completed Subjects: Because subjects served as their own control, both groups included together.
Arm/Group | All Completed Subjects
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04553913/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT04553913/ICF_001.pdf